CLINICAL TRIAL: NCT04417660
Title: A Phase II, Open-Label Trial of Bintrafusp Alfa (M7824) in Subjects With Thymoma and Thymic Carcinoma
Brief Title: Bintrafusp Alfa (M7824) in Subjects With Thymoma and Thymic Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200097; 20-C-0097
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Thymic Epithelial Tumor; Recurrent Thymoma; Thymic Cancer
Keywords: Thymoma; thymic cancer; Immune Checkpoint Inhibition; programmed death ligand 1 (PD-L1)
MeSH Terms: conditions — Thymic epithelial tumor; Thymoma; Thymus Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bintrafusp alfa (M7824) (Experimental): Bintrafusp alfa will be administered at a dose of 1200 mg intravenously once every two weeks until disease progression or development of intolerable adverse events.
  Interventions: Drug: M7824

INTERVENTIONS:
Drug: M7824 — Bintrafusp alfa will be administered at a dose of 1200 mg intravenously once every two weeks until disease progression or development of intolerable adverse events.

SUMMARY:
Background:

Thymoma and thymic carcinoma are diseases of the thymus. Platinum-based chemotherapy is the standard treatment for these diseases. But in many cases, the disease returns after treatment. Researchers want to see if a new drug can help.

Objective:

To see if bintrafusp alfa (M7824) is an effective treatment for thymoma and thymic carcinoma.

Eligibility:

People age 18 and older who have thymoma or thymic cancer and their disease returned or progressed after treatment with at least one platinum-containing chemotherapy treatment plan.

Design:

Participants will be screened under a separate protocol. Their medical, medicine, and treatment history will be reviewed. They will have a tumor biopsy if they do not have a sample.

Participants will get the study drug once every 2 weeks as an intravenous infusion. For this, a small plastic tube is put into an arm vein.

During the study, participants will undergo the following:

Medicine review

Physical exam

Review of their symptoms and their ability to perform their normal activities

Blood and urine tests

Thigh muscle scan (using MRI)

Tumor assessment (using MRI or CT)

Heart and lung function tests

Thyroid gland test

Skin assessment.

Participants may have tumor biopsies. Some of their blood and biopsy samples will be used for gene testing.

Participants may take the study drug until their disease worsens or they cannot tolerate treatment.

Participants will have follow-up visits 2 and 6 weeks after stopping treatment. Then they will have long-term follow-up visits every 3 months. These may include imaging scans. Visits may be done by phone, with scans (if needed) done at their doctor s office.

DETAILED DESCRIPTION:
Background

Platinum-based chemotherapy is the standard of care for advanced unresectable thymic epithelial tumors (TETs). However more than half of these patients experience disease recurrence and require second-line therapy.

There are no approved drugs for treatment of recurrent thymoma and thymic carcinoma and new therapeutic options are needed for patients who have disease progression on or after platinum-containing therapy.

We have demonstrated the safety and clinical activity of immune checkpoint inhibition in patients with recurrent TETs. In an ongoing trial (NCT03076554) we have shown that avelumab, an anti-programmed death ligand-1 (PD-L1) antibody, induces major responses and has an acceptable safety profile.

Combination immunotherapy is under evaluation for treatment of various cancers but has not been studied for the treatment of TETs. Immunotherapy targeting the PD-1/PD-L1 axis can be combined with other immune checkpoint inhibitors, cancer vaccines and anti-cytokine therapy.

Bintrafusp alfa, a bifunctional fusion protein that targets PD-L1 and transforming growth factor-Beta (TGF-Beta) has shown activity against heavily pre-treated solid tumors including non-small cell lung cancer previously treated with single-agent anti-PD-1/PD-L1 inhibitors.

Retrospective analysis of pre-chemotherapy tissue obtained from 20 patients with stage IV thymic carcinoma and 13 cases of stage III/IV thymoma, showed TGF-Beta expression in 65% cases of thymic carcinoma and 15% cases of thymoma with a lower median survival among patients with thymic carcinoma (30 months versus 63 months).

As part of a phase I clinical trial, treatment with bintrafusp alfa resulted in a brief period of disease stabilization and no immune-related adverse events in one patient with heavily pre-treated, WHO subtype B3 thymoma with a large disease burden

Further investigation of Bintrafusp alfa in patients with recurrent TETs is needed to define the clinical activity and safety of this drug in patients with TETs.

Primary Objectives

To determine the objective response rate (ORR) to bintrafusp alfa in participants with relapsed or refractory thymoma and thymic carcinoma.

Eligibility

Participants >= age 18 years with histologically confirmed, unresectable thymoma or thymic carcinoma who have previously been treated with at least one platinum-containing chemotherapy regimen with progressive disease prior to study entry.

Progressive and measurable disease prior to enrollment

No history of autoimmune disease, with exception of vitiligo, autoimmune thyroid disease, or pure red cell aplasia that are adequately managed with medical therapy

Adequate renal, hepatic and hematopoietic function

Design

This will be a single-arm, phase II study to determine the clinical activity of treatment with Bintrafusp alfa in participants with relapsed or refractory thymoma and thymic carcinoma.

Bintrafusp alfa will be administered at a dose of 1200 mg intravenously once every two weeks until disease progression or development of intolerable adverse events. The two-week period will constitute one cycle.

A Simon optimal two-stage phase II trial design will be used to rule out unacceptably low response rate of 20% in favor of an improved response rate of 45%

Participants will be enrolled in 2 disease cohorts, thymoma and thymic carcinoma, with up to 17 evaluable participants of each tumor type. Accrual ceiling will be set at 44 participants to account for inevaluable participants and screen failures.

Participants who have completed 12 months of treatment with an ongoing response or disease stability (for >= 6 months) will be given an option of discontinuing active treatment with the ability to reinstitute treatment on one occasion if radiological or clinical disease activity is noted during follow-up. All eligibility criteria should be met at the time of restarting treatment with bintrafusp alfa.

Tumor response will be assessed after completion of every third cycle (6 weeks) using modified immune-related RECIST criteria. When possible, an optional tumor biopsy will be conducted pre-treatment, after 3 doses in participants responding to treatment or at 6 weeks, whichever is sooner, to evaluate treatment-related, intra-tumoral changes.

Exploratory objectives include immune correlative studies to analyze immune cell subsets, PD-L1 expression and evaluation of soluble factors and intra-tumoral changes before and after bintrafusp alfa treatment.

ELIGIBILITY:
* IINCLUSION CRITERIA:
* Participants must have histologically confirmed (by the pathology department/CCR/NCI) thymoma or thymic carcinoma.
* Participants must have had at least one prior line of platinum-based chemotherapy. Progressive disease must be documented prior to study entry and participants must have advanced, unresectable disease that is not amenable to surgical resection.
* Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST1.1.
* Participants must be aged >=18 years.
* ECOG performance status <=1.
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count: >= 1,500/mm3 OR >= 1.5 x 10(9)/L
  * platelets: >=> 100,000/mm3 OR >= 100 x 10(9)/L
  * hemoglobin: >= 9g/dL (may have been transfused)
  * total bilirubin: <= the upper limit of normal range (ULN) OR <= 3.0 x ULN for participants with documented metastatic disease to the liver
  * AST(SGOT)/ALT(SGPT): <= 1.5 x ULN OR <= 5 x ULN for participants with documented metastatic disease to the liver
  * ALP: <= 2.5 x ULN
  * creatinine clearance: >= 60 mL/min/1.73 m2 calculated by calculated using eGRF in the clinical lab
  * INR: normal INR, per institutional guidelines
  * PT: <= 1.5 x ULN
  * aPTT: <= 1.5 x ULN
* Negative serum or urine pregnancy test at screening for individuals of childbearing potential (IOCBP). NOTE: IOCBP is defined as any individual who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. If necessary, to confirm postmenopausal status an FSH level will be included at screening. The effects of Bintrafusp alfa on the developing human fetus are unknown. For this reason, individuals of childbearing potential and those that can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for at least 2 months after the last dose of the drug.
* Participants with previously treated brain or CNS metastases are eligible provided that the participant has recovered from any acute side effects of radiotherapy and does not require treatment with steroids, and any whole brain radiation therapy was completed at least 2 weeks prior to enrollment.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bintrafusp alfa.
* History of anaphylaxis or recent (within 5 months) history of uncontrollable asthma.
* Prior treatment with PD-1 or PD-L1-directed immune checkpoint blockade is not permitted. Prior treatment with other immunomodulating drugs such as cancer vaccines is permitted based on investigators discretion as long as treatment was not discontinued due to life-threatening adverse events (laboratory abnormalities alone with prior therapy will not exclude participants from this trial).
* Concurrent treatment with a non-permitted drug
* Prior anticancer treatment within 14 days before treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative bone directed radiotherapy], immune therapy, or cytokine therapy except for erythropoietin); major surgery within 14 days before treatment (excluding prior diagnostic biopsy); prior systemic therapy (or 5 half-lives of a drug, whichever is shorter) with immunosuppressive agents within 14 days before treatment; use of hormonal agents for anti-cancer therapy within 7 days before treatment; or use of any investigational drug within 14 days before treatment.

Note: Participants receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before treatment.

* History of previous malignant disease within the last 3 years with the following exceptions: basal or squamous cell carcinoma in situ of the skin treated with curative intent, endoscopically resected GI cancers limited to the mucosal layer without recurrence in > 1 year, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary or follicular thyroid carcinoma, and superficial/non-muscle invasive bladder cancer.
* Active brain or CNS metastases causing clinical symptoms or metastases that require therapeutic intervention.
* Active or history of autoimmune disease that might deteriorate when receiving an immune-stimulatory agent, with the exception of diabetes type I, vitiligo, psoriasis, autoimmune thyroid disease not requiring immunosuppressive treatment, or pure red cell aplasia that are adequately managed with medical therapy. In addition, anti-acetylcholine receptor binding antibodies will be checked during screening and participants will be ineligible if results are positive, even if there is no clinical history of autoimmune disease.
* Participants receiving systemic corticosteroids at doses > 10 mg daily prednisone equivalent will be excluded. However, participants on inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of autoimmune disease
* Active infection requiring systemic therapy or significant acute or chronic infections including, among others:

  * Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
  * Known history of testing positive for HIV or testing positive for HIV at screening or known acquired immunodeficiency syndrome.

HIV-positive TET participants are ineligible because of the risk of developing opportunistic infections after treatment with an immune checkpoint inhibitor. Additionally, TET participants are at higher risk of developing opportunistic infections due to underlying immune defects. Prior cases of disseminated herpes virus, cytomegalovirus and fungal infections have been documented in this patient population.

* Prior organ transplantation including allogenic stem-cell transplantation, Participants who have had prior transplants that do not require immunosuppression are eligible.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 5 Grade > 1); however, alopecia, sensory neuropathy Grade <= 2, or other Grade <= 2 not constituting a safety risk based on investigator s judgment are acceptable.
* Participants unwilling to accept blood products as medically indicated.
* Pregnant or lactating individuals. Pregnant individuals are excluded from this study because Bintrafusp alfa is in the class of agents known as antineoplastics/monoclonal antibodies with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Bintrafusp alfa, breastfeeding should be discontinued if the mother is treated with Bintrafusp alfa.
* Known alcohol or drug abuse.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cerebral vascular accident/stroke < 6 months prior to enrollment, myocardial infarction < 6 months prior to enrollment, or psychiatric illness/social situations that would limit compliance with study requirements. All other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, drug-induced pneumonitis requiring oral or IV steroids, interstitial lung disease, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study. Participants with history of bleeding diathesis or recent major bleeding events considered by the Investigator as high risk for investigational drug treatment are also excluded.
* Administration of live vaccine within 4 weeks prior to treatment, with the exception of vaccination against COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | from the start of the treatment until disease progression/recurrence
  overall response rate for M7824 based on RECIST criteria

SECONDARY OUTCOMES:
Duration of response, progression free survival & overall survival | from the start of the treatment until disease progression/recurrence
  To determine duration of response, progression free survival and overall survival in participants with recurrent thymic epithelial TETs
Safety & tolerability of M7824 | from the start of the treatment until disease progression/recurrence
  To determine the safety and tolerability of 1200 mg M7824 administered once every 2 weeks in participants with thymoma and thymic carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Remon J, Girard N, Novello S, de Castro J, Bigay-Game L, Bernabe R, Greillier L, Mosquera J, Cousin S, Juan O, Sampayo M, Besse B. PECATI: A Multicentric, Open-Label, Single-Arm Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab and Lenvatinib in Pretreated B3-Thymoma and Thymic Carcinoma Patients. Clin Lung Cancer. 2022 May;23(3):e243-e246. doi: 10.1016/j.cllc.2021.07.008. Epub 2021 Jul 20. PMID 34393061
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0097.html